CLINICAL TRIAL: NCT07278557
Title: Assessment of Sparing Parotid Ducts Via MRI Sialography for Reduced Patient-Reported Xerostomia Following Radiotherapy for Oropharynx Cancer
Brief Title: Sparing Parotid Ducts Via MRI Sialography for Reduced Patient-Reported Xerostomia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LCCC2444; UG3DE033389 (NIH)
Record Dates: First submitted 2025-12-03; First posted 2025-12-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer
Keywords: Radiation-induced xerostomia; parotid gland dose; radiation dose; parotd sparing; MRI sialography
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: This study is double-masked, ensuring that both treating physicians and study participants are masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Participants randomized to this arm will have their organs-at-risk include the expanded parotid ducts. Treatment planning will aim to explicitly minimize the dose to these structures. If achieving this dose is not possible, it will be documented as a study deviation, but treatment will proceed.
  Interventions: Device: MRI sialography; Other: Parotid Duct Sparing Radiation Therapy Planning
- Standard Arm (Active Comparator): Participants in this arm will undergo treatment planning using the overall parotid gland volume as the organ-at-risk, following the standard clinical practice. Entire parotid gland will be considered, not the parotid ducts.
  Interventions: Device: MRI sialography; Other: Parotid Sparing Radiation Therapy Planning

INTERVENTIONS:
Device: MRI sialography — Prior to radiation therapy treatment planning, all participants will undergo magnetic resonance imaging (MRI) sialography in order to visualize patients' parotid ducts. This will enable these organs-at-risk to be spared during radiation treatment planning
Other: Parotid Duct Sparing Radiation Therapy Planning — Radiation therapy will be administered based on treatment planning that aims to minimize the dose to the parotid ducts.
  Arms: Experimental Arm
Other: Parotid Sparing Radiation Therapy Planning — Radiation therapy will be administered based on treatment planning that uses the entire parotid gland volume as the organ-at-risk, in accordance with standard clinical practice. The parotid ducts will not be considered separately.
  Arms: Standard Arm

SUMMARY:
Radiation-induced xerostomia (dry mouth) is one of the most common and severe side effects for patients receiving radiation therapy for head and neck cancer. New approaches are needed to reduce this side effect and improve patients' quality of life after treatment.

This is a Phase II, single-center, double-masked, parallel-arm, randomized controlled trial. It compares MRI-guided parotid ductal sparing to the standard approach of mean parotid gland sparing, focusing on patient-reported dry mouth outcomes in individuals receiving definitive radiotherapy for oropharyngeal cancer.

DETAILED DESCRIPTION:
Radiation-induced dry mouth (xerostomia) is the most commonly reported long-term side effect in patients receiving radiation therapy (RT) for head and neck cancer. It occurs when saliva production decreases and the saliva becomes thicker. Patients with xerostomia often have trouble chewing, swallowing, and speaking, and are more likely to develop tooth decay. These problems can significantly lower a patient's quality of life-and the impact tends to get worse over time.

The most common way to reduce radiation-related dry mouth is by limiting the average radiation dose to the parotid glands (which produce saliva). However, this is often not possible because of the patient's anatomy, and many patients still report moderate to severe symptoms long after treatment.

To reduce side effects, some studies have tested giving a lower radiation dose (60Gy instead of the usual 70Gy) in patients with low-risk, HPV-associated tumors. While this has helped improve overall symptoms, xerostomia still remains the most severe and persistent problem reported by patients.

New strategies are needed to better protect patients from radiation-related dry mouth and help maintain their quality of life after treatment. Recent research shows that the parotid gland does not respond evenly to radiation; certain areas, especially large salivary ducts where stem/progenitor cells live, may be key for recovery after damage. If these ducts can be located during treatment planning, the radiation dose to them could be reduced.

A pilot study showed that using MRI sialography to identify the parotid ducts and plan radiation therapy around them is both possible and promising. Patients who received this type of duct-sparing RT had fewer moderate-to-severe dry mouth symptoms compared to patients treated with standard RT (46% vs. 71% at 6 months, and 36% vs. 50% at 12 months post-treatment).

A larger, randomized study is still needed to confirm whether reducing radiation dose to the parotid ducts can meaningfully lower the risk of xerostomia and improve recovery after radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

To participate in this study a subject must meet all of the eligibility criteria outlined below. Eligibility must be maintained for the subject to be considered eligible for ongoing trial participation.

* Provide written informed consent to participate in the study and HIPAA authorization for release of personal health information.
* Able to comply with study procedures based on the judgment of the clinical investigator.
* Male or female, aged ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group performance status 0-2 at the time of consent.
* Women of reproductive potential must use highly effective contraception.
* T0-4, N0-3, M0 stage cancer of the oropharynx (American Joint Committee on Cancer Staging System 8th edition) planned for definitive radiotherapy +/- chemotherapy.
* No contraindications for magnetic resonance imaging (MRI).

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation

In this study:

* Patients with Sjogren's disease or baseline xerostomia.
* Patients with lesions involving the salivary glands on diagnostic imaging
* Patients with an allergy to lemon juice
* Prior lifetime history of radiation therapy to the head and neck
* Current pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
The rate of xerostomia score based on the University of Michigan Xerostomia -6 months Questionnaire - 6 months | 6 months
  The rate of xerostomia score based on the University of Michigan Xerostomia Questionnaire (UMXQ) will be determined. UMXQ is an eight-item patient-reported instrument designed to assess the severity of xerostomia (dry mouth), gauging symptoms both during and outside of eating or chewing. The score ranges from 0 to 100, with higher scores indicating worse xerostomia. Participants treated with parotid ductal sparing radiotherapy will be compared.

SECONDARY OUTCOMES:
Salivary flow unstimulated | at 6 and 12 months
  Participants will be asked not to eat, drink (except water), or smoke for at least one hour before the test and will rinse their mouth with deionized water five minutes prior to collection.
  Participants will sit comfortably with their head slightly forward and allow saliva to naturally accumulate in the mouth. They will spit into a pre-weighed cup every 60 seconds for five minutes. After a five-minute rest, stimulated saliva will be collected. Participants will chew paraffin gum for one minute at a controlled rate, then continue chewing and spit accumulated saliva into a separate pre-weighed cup every 60 seconds for five minutes.
Salivary flow stimulated | at 6 and 12 months
  Stimulated saliva will be collected five-minute rest after the unstimulated saliva collection. Participants will chew paraffin gum for one minute at a controlled rate, then continue chewing and spit accumulated saliva into a separate pre-weighed cup every 60 seconds for five minutes.
The rate of xerostomia score based on the University of Michigan Xerostomia Questionnaire- 12 months | 12 months
  The rate of xerostomia score based on the University of Michigan Xerostomia Questionnaire (UMXQ) will be determined. UMXQ is an eight-item patient-reported instrument designed to assess the severity of xerostomia (dry mouth), gauging symptoms both during and outside of eating or chewing. The score ranges from 0 to 100, with higher scores indicating worse xerostomia. Participants treated with parotid ductal sparing radiotherapy will be compared.
The rate of xerostomia score based on the MD Anderson Symptom Inventory Head and Neck (MDASI - HN)- 12 months | 12 months
  The rate of xerostomia will be assessed using the MD Anderson Symptom Inventory-Head and Neck (MDASI-HN), a validated patient-reported outcome measure evaluating symptom severity and impact on daily functioning in head and neck cancer patients. It includes 13 core symptom items (e.g., fatigue, pain, nausea), 9 head and neck-specific items (e.g., swallowing difficulty, dry mouth, taste changes, voice problems), and 6 interference items assessing effects on mood, work, and enjoyment of life. Each item is rated on a 0-10 scale, where 0 indicates no symptom or interference and 10 indicates the worst severity or complete interference. Scores are calculated as the mean of core symptom items for total severity, the mean of head and neck-specific items, and the mean of interference items.

CONTACTS AND LOCATIONS:
Overall Officials: David Fried, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared with other researchers per the NIHs data management and sharing policy.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials